CLINICAL TRIAL: NCT06921720
Title: ATP (Adenosine Triphosphate) Concentration Measurement by Phosphorus-31 Spectroscopy in Phosphate Diabetes
Brief Title: Phosphorus-31 Spectroscopy in Phosphate Diabetes
Acronym: Phos-ATP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL24_0352; 2024-A02748-39 (Other: ID-RCB)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Phosphate Diabetes; X-linked Hypophosphatemia
Keywords: Hypophosphatemia; XLH; phosphate diabetes; muscle; 31P-MRS
MeSH Terms: conditions — Hypophosphatemia, Familial; Familial Hypophosphatemic Rickets; Hypophosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with phosphate diabetes (Experimental): patient aged ≥ 10 years with phosphate diabetes, meaning genetically confirmed XLH or phosphate diabetes of another origin characterized by hypophosphatemia with a decreased Tm (tubular maximum) /GFR (glomerular filtration rate).
  Interventions: Diagnostic Test: intra-muscular ATP values in phosphate diabetes; Diagnostic Test: intra-muscular phosphate values in phosphate diabetes
- Pediatric and adult controls (Experimental): Pediatric patients aged 10 to 17 years without chronic kidney disease, without hypophosphatemia, without muscle abnormalities, matched for age and sex.
  Adult control patient without chronic kidney disease, without hypophosphatemia, without muscle abnormalities, without malnutrition, and matched for age and sex.
  Interventions: Diagnostic Test: intra-muscular ATP values in phosphate diabetes; Diagnostic Test: intra-muscular phosphate values in phosphate diabetes

INTERVENTIONS:
Diagnostic Test: intra-muscular ATP values in phosphate diabetes — intra-muscular ATP values [ATPi] (measured by 31P-MRS / Phosphorus-31 nuclear magnetic resonance) at rest and during standardized exercise in patients with phosphate diabetes.
Diagnostic Test: intra-muscular phosphate values in phosphate diabetes — intra-muscular phosphate values (measured by 31P-MRS) at rest and during standardized exercise in patients with phosphate diabetes.

SUMMARY:
Phosphate diabetes is defined by urinary phosphate wasting due to impaired tubular reabsorption. It can be classified based on either a genetic or acquired origin. Chronic hypophosphatemia causes rickets in children, leading to growth disorders, bone deformities, and bone pain. In adults, it results in osteomalacia, pseudofractures, as well as muscle fatigue and weakness during exertion.

X-linked hypophosphatemia (XLH) is a common cause of hereditary rickets linked to renal phosphate loss due to elevated FGF23 levels, most often caused by mutations in the PHEX (Phosphate Regulating Endopeptidase X-Linked) gene. Clinical trials have already demonstrated significant improvements in the quality of life of patients with XLH following the approval of the anti-FGF23 antibody, Burosumab.

However, there are other causes of phosphate diabetes, such as tumor-induced osteomalacia (TIO), proximal tubulopathies (Dent disease, cystinosis), or mutations in Npt2a/C.

As described above, patients with phosphate diabetes report bone pain and variable muscle fatigue depending on the underlying cause. These symptoms can significantly impact quality of life by limiting physical activities early on. However, standard quality-of-life questionnaires often lack the specificity to accurately assess these symptom-related impairments. At present, the investigators lack objective biomarkers that can quantitatively assess subclinical metabolic abnormalities at the muscular level in these patients.

Various data from animal models and preclinical studies suggest direct links between serum phosphate levels, intracellular phosphate (Pi), ATP production, and altered muscle metabolism. Muscle tissue requires energy, primarily derived from ATP hydrolysis. ATP is synthesized via mitochondrial oxidative phosphorylation, which is regulated by intracellular phosphate levels.

In five XLH patients, older studies compared intracellular Pi levels to those of five healthy controls and showed a decrease in Pi without a change in intracellular ATP. Smith et al. found ATP concentrations within the lower limit of normal at rest, while Pesta et al. reported a decrease in muscle ATP concentration in hypophosphatemic mice, which normalized after correcting serum phosphate levels.

Two recent studies using 31-phosphorus magnetic resonance spectroscopy (31P-MRS) showed no change in intracellular ATP levels in XLH patients, both before muscle activity and after burosumab treatment. However, these studies were conducted at rest. Yet, the main issue for patients lies in physical activity, as quality-of-life impairments often begin with limitations in daily physical tasks. Moreover, no current data are available on intracellular Pi or ATP levels in other forms of phosphate diabetes.

These parameters can be measured in vivo, non-invasively, using 31P-MRS. This technique employs a standard 3T MRI scanner equipped with a multinuclear coil to detect phosphorus instead of protons. It allows for ATP, Pi, and phosphocreatine concentrations to be measured every 2 minutes and 45 seconds. The procedure is non-irradiating, requires no contrast injection, and focuses on the patient's leg, meaning the whole body does not need to be inside the MRI scanner.

Additionally, in FGF23-mediated phosphate diabetes, calcitriol suppression leads to renin-angiotensin-aldosterone system (RAAS) activation and hypertension. In contrast, proximal tubulopathies cause salt wasting. The third sodium compartment (non-osmotically active sodium stored in subcutaneous and muscle tissue) can be assessed non-invasively using 23Na-MRI (sodium-23 MRI), which also uses a 3T (3 tesla) MRI scanner and a multinuclear coil to detect sodium signals under the same conditions as 31P-MRS.

Patients with XLH also exhibit a distinct metabolic profile, with an increased risk of obesity, hypertension, left ventricular hypertrophy, and elevated uric acid levels.

The goal of the study is to quantitatively measure intramuscular ATP, intracellular phosphate (Pi), intracellular pH, and phosphocreatine both before and during exercise in patients with phosphate diabetes. The study also aims to characterize the mitochondrial and metabolic profile of these patients and assess the non-osmotically active third sodium compartment in these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Patients:
* Patient ≥ 10 years old with phosphate diabetes, i.e., genetically confirmed XLH or phosphate diabetes of another origin characterized by hypophosphatemia with a decreased Tm/GFR.
* Patient has given consent to participate in the study.
* Signed consent (by both legal representatives for minor patients).
* Patient regularly followed up within the pediatric nephrology services at the Femme Mère Enfant hospital and the nephrology-functional exploration services at the Edouard Herriot hospital.

Inclusion Criteria for Pediatric Controls:

* Patient aged 10 to 17 years, without chronic kidney disease, without hypophosphatemia, without muscular abnormalities, and without growth disorders.
* Patient has given consent to participate in the study.
* Signed consent (by both legal representatives for minor patients).
* Patient regularly followed up within the pediatric nephrology services at the Femme Mère Enfant hospital.

Inclusion Criteria for Adult Controls:

* Patient without chronic kidney disease, without hypophosphatemia, without muscular abnormalities, and without malnutrition.
* Patient has given consent to participate in the study.
* Signed consent.
* Patient regularly followed up within the renal functional exploration services at the Edouard Herriot hospital.

Exclusion Criteria:

* Pregnant, parturient, or breastfeeding women
* Individuals deprived of liberty by a judicial or administrative decision
* Individuals receiving psychiatric care
* Individuals admitted to a healthcare or social institution for purposes other than research
* Adults under legal protection (guardianship, curators)
* Individuals not affiliated with a social security system or benefiting from a similar scheme
* Subjects participating in another interventional study with an exclusion period still in effect at pre-inclusion
* General contraindications for MRI: wearing a pacemaker/ICD (implantable cardiac device) or mechanical heart valves not MRI-compatible, presence of non-MRI-compatible equipment, presence of metallic objects.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference in intra-muscular ATP values [ATPi] (measured by 31P-MRS) at rest and during standardized exercise in patients with phosphate diabetes. | At rest and during Brief physical exercise of foot flexion/extension to fatigue using a calibrated elastic band within the MRI (Magnetic resonance imaging). For patients with Burosumab on day 7 after the injection."
  measured on the calf

SECONDARY OUTCOMES:
Difference in intra-muscular phosphate values (measured by 31P-MRS) at rest and during standardized exercise in patients with phosphate diabetes. | At rest and during Brief physical exercise of foot flexion/extension to fatigue using a calibrated elastic band within the MRI. For patients with Burosumab on day 7 after the injection
  measured on the calf
Absolute values of ATPi and Pi (31P-MRS) before and during standardized exercise in patients with phosphate diabetes compared to age-matched control subjects, in patients with XLH compared to other types of phosphate diabetes matched for age, in patients | At rest and during Brief physical exercise of foot flexion/extension to fatigue using a calibrated elastic band within the MRI. For patients with Burosumab on day 7 after the injection.
  measured on the calf
Correlation between absolute values of ATPi and Pi (31P-MRS) at rest and during standardized exercise in patients with phosphate diabetes and the following outcomes | At rest and during Brief physical exercise of foot flexion/extension to fatigue using a calibrated elastic band within the MRI. For patients with Burosumab on day 7 after the injection.
  Correlation between absolute values of ATPi and Pi (31P-MRS) at rest and during standardized exercise in patients with phosphate diabetes and the following outcomes:6-minute walk test, Maximal VO2 (rate (V) of oxygen (O₂)), Quality of life scale, Mitochondrial and metabolic profile of PBMCs (peripheral blood mononuclear cell) Quality of life scale: SF36 (36-Item Short Form Survey), WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index), BPI-SF (Brief Pain Inventory - Short Form) et BFI (big five inventory) PED (pediatric) SCALE, test Sports and physical functioning

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital femme mère enfant, hospices civils de Lyon, Bron
  - Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon